CLINICAL TRIAL: NCT05389085
Title: Fast Track Diagnosis of Malignant Melanoma by Two Advanced Imaging Technologies and Tumour Tapestripping of RNA and Lipids
Brief Title: Fast Track Diagnosis of Skin Cancer by Advanced Imaging Technologies and Tumour Tapestripping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Mette Mogensen, Assoc. Prof, Chief Consultant, MD, PhD, University Hospital Bispebjerg and Frederiksberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2200972
Record Dates: First submitted 2022-04-28; First posted 2022-05-24 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Skin Cancer; Malignant Melanoma
Keywords: diagnostic imaging; pigmented skin neoplasm; tape-stripping; photoacoustic techniques; confocal microscopy
MeSH Terms: conditions — Skin Neoplasms; Melanoma | interventions — Erythrocyte Volume

STUDY DESIGN:
Intervention Model Description: This prospective non-blinded clinical study will include 75 patients with suspicious pigmented skin tumours (i.e. malignant melanomas, lentigo maligna, pigmented nevi, and pigmented basal cell carcinomas) referred to or diagnosed at Dept. of Dermatology, BFH. All tumours are histologically verified by skin biopsy or surgical excision. Patients who meet the inclusion criteria will be enrolled if they consent. If patients demonstrate more than one skin tumour within the same anatomical location, only one lesions will be included and scanned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective non-blinded clinical study (Other): All patients enrolled with with suspicious pigmented skin tumours will be scanned with reflectance confocal microscopy and photoacoustic imaging by an experienced examiner in a 30 minutes to 1-hour session. Subsequently, material for RNA and lipid analysis is obtained from tape-stripped lesional skin at the bedside. The skin tumors in patients enrolled will subsequently be treated according to hospital and national guidelines.
  Interventions: Diagnostic Test: Reflectance confocal microscopy (RCM), Photoacoustic imaging (PAI) and tape-strippng of RNA and lipids

INTERVENTIONS:
Diagnostic Test: Reflectance confocal microscopy (RCM), Photoacoustic imaging (PAI) and tape-strippng of RNA and lipids — In vivo RCM will be used to diagnose pigmented tumours at a cellular level and provide information on skin microarchitecture. MSOT detects skin chromophores as melanin, hemoglobin, water, collagen, and lipids, which will be included in analysis of diagnostic accuracies. MSOT will also be used to measure tumour thickness; delineate tumour borders and analyze blood flow in blood vessels. Potential diagnostic features from each lesion type will be tested. RNA and lipid profiles from tape stripping results will be compared to imaging and histopathology diagnosis.
  Other Names: Vivascope Multilaser 1500®, Vivascope GmbH, Munich, Germany, https://www.vivascope.de/medical-imaging/ and provided in Denmark by Scan-Med A/S, Dalgårdsvej 17, 8220 Brabrand.; MSOT Acuity from iThera Medical GmbH, Munich, Germany, https://www.ithera-medical.com/technology/ not sold in Denmark but provided directly from the company.

SUMMARY:
In this clinical feasibility study the investigators will test and compare two advanced optical imaging technologies, lipid and RNA tape stripping with regards to diagnostic accuracies for fast bedside diagnosis of pigmented skin tumours.

DETAILED DESCRIPTION:
This original clinical research project utilizes cutting-edge medical imaging technologies for diagnosis of pigmented skin tumours, combined for the first time in Denmark, with molecular RNA and lipid analysis of superficial tumours cells. The scanning technologies are reflectance confocal microscopy (RCM), which is a microscope applied directly to the skin surface, and photoacoustic imaging, also termed multispectral optoacoustic imaging (MSOT), which is an imaging technology actually listening to the skin for immediate bedside diagnosis of pigmented skin tumors. The hypothesis is that treatment guided by diagnostic bedside skin scanning, combined with tumour tape-stripping and RNA and lipid analysis can increase diagnostic accuracy compared to visual inspection of the skin tumour and thus decrease time delay from diagnosis to efficient treatment

ELIGIBILITY:
Inclusion Criteria:

1. 75 patients with histologically verified pigmented skin tumours on areas of the body where scanning is feasible with both imaging systems
2. Patients with clinically suspicious skin tumours, that are not yet biopsied, if the patient is willing to undergo a skin biopsy from the suspicious lesion
3. > 18 years of age at baseline
4. Legally competent, able to give verbal and written consent
5. Communicate in Danish verbally as well as in writing
6. Subject in good general health, is willing to participate and able to give informed consent and can comply with protocol requirements.

Exclusion Criteria:

1. Individuals with other skin diseases in the skin area of interest
2. Individuals who´s skin tumour is not accessible for imaging e.g. inside the ear, inside nostrils, on eyelids
3. Subjects who will not undergo a skin biopsy after imaging of the suspicious skin tumour and who have not had a skin biopsy taken from the tumour prior to referral
4. Pregnancy
5. Women of child-bearing potential not using a contraceptive agent at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy. The primary objective i to test and compare two advanced optical imaging technologies, lipid and RNA tape stripping with regards to diagnostic accuracies for fast bedside diagnosis of pigmented skin tumours. | All patients will be scanned by an experienced examiner in a 30 minutes to 1 hour session.
  Will be presented as sensitivity, specificity, and positive and negative predictive values. Tumor thickness measurements using MSOT will be measured and reported in millimeters. The blood flow in dermal blood vessels will be measured quantitatively by MSOT and vascular morphology will be described qualitatively. RCM images will be evaluated qualitatively regarding cellular changes, skin micromorphology and characteristic malignant melanoma features.

SECONDARY OUTCOMES:
Analysis of RNA molecules of surface cells from tape stripping | Up to 6 months
  Examination of the expression of a total of 22 selected RNA molecules in suspicious skin tumours will be investigated by quantitative reverse-transcription methods with the use of the TaqMan method (Thermo Fisher Scientific).
Lipid analysis from tape-stripping | Up to 6 months
  We will analyze lipids obtained by tape-stripping from surface cells in pigmented lesions by ex vivo spectroscopic near-infrared optical coherence tomography (OCT), performed at DTU: Dept of Photonics Lab Facilities.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Mogensen, MD, PhD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Dept of Dermatology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
The study will be performed in accordance with ICH GCP Guidelines and Danish Health care authorities. It will be registered at The National Committee on Health Research Ethics, Danish Medicines Agency, and The Danish Data Protection Agency. Study conduction and reports are in accordance with GCP CPMP/ICH/135/95 and European Medicines Agency directive 2001/83/EC.
  The study will be published in an international dermatological journal and presented at scientific conferences. Positive, negative and inconclusive results will be published and inconclusive results will be published at www.clinicaltrials.gov and www.clinicaltrialsregister.eu . Authorships are given according to the Vancouver guidelines.